CLINICAL TRIAL: NCT03045354
Title: The Effect of Carbohydrate-Containing Foods at Breakfast on Food Intake, Glycemic Response, and Subjective Appetite in Normal Weight and Overweight/Obese Children
Brief Title: Dietary Carbohydrate Consumption at Breakfast on Food Intake, Glycemic Response, and Subjective Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Nick Bellissimo, Associate Professor, School of Nutrition, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: REB2016-227
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Childhood Obesity; Breakfast
Keywords: children; dietary carbohydrates; satiety; appetite; blood glucose; solanum tuberosum; obesity; breakfast
MeSH Terms: conditions — Pediatric Obesity; Obesity | interventions — lunatusin, Phaseolus lunatus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Mashed potatoes (Experimental): Eggs with a side of mashed potatoes
  Interventions: Other: Mashed potatoes
- French fries (Experimental): Eggs with a side of French fries
  Interventions: Other: French fries
- Beans (Experimental): Eggs with a side of beans
  Interventions: Other: Beans
- Traditional breakfast (Experimental): Cereal, milk, toast and jam
  Interventions: Other: Traditional breakfast
- Breakfast skipping (Experimental): No breakfast
  Interventions: Other: Breakfast skipping

INTERVENTIONS:
Other: Mashed potatoes — Isocaloric (450 kcal) breakfast treatments of eggs with a side of mashed potatoes
  Arms: Mashed potatoes
Other: Traditional breakfast — Isocaloric (450 kcal) control breakfast treatments of cereal, milk, toast and jam
  Arms: Traditional breakfast
Other: Breakfast skipping — No breakfast
  Arms: Breakfast skipping
Other: French fries — Isocaloric (450 kcal) breakfast treatments of eggs with a side of French fries
  Arms: French fries
Other: Beans — Isocaloric (450 kcal) breakfast treatments of eggs with a side of beans
  Arms: Beans

SUMMARY:
The purpose of this study is to determine the effect of carbohydrates of familiar breakfast meals on glycemic response, subjective appetite, and food intake in normal weight (NW) and overweight or obese (OW/OB) children.

DETAILED DESCRIPTION:
Regular breakfast eating NW and OW/OB children, 9-14 years of age, will participate in the experiment. Four isocaloric (450 kcal) breakfasts (eggs with a side of French fries, mashed potatoes, or beans, and control breakfast of milk, cereal and toast) and breakfast skipping will be examined. On five separate mornings, 7 days apart and after a 12 hour overnight fast, each participant will receive one of the four breakfasts or skip breakfast, in a randomized counterbalanced order. Participants will be given an ad libitum lunch 3 hours after breakfast and parents will report the rest of day food record for food intake analysis. Blood glucose will be measured via finger-prick at baseline, and 30, 60, 120, and 180 minutes after breakfast consumption. Subjective appetite will be measured with a visual analogue scale at baseline and every 15 minutes for 1 hour, and every hour for 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* be between 9 and 14 years of age
* be healthy, and have been born at term
* not be taking any medications
* not have allergies or sensitivities to potatoes, eggs, gluten, dairy, or beans
* NW (between the 5th and 85th BMI percentile for age and gender)
* OW/OB (>85th BMI percentile for age and gender)

Exclusion Criteria:

* food sensitivities, allergies, or dietary restrictions
* health, learning, emotional, or behavioural problems
* receiving any medications

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Short-term food intake (kcal) | 3 hours after breakfast
  Participants will consume an ad libitum lunch 3 hours post breakfast consumption.

SECONDARY OUTCOMES:
Subjective appetite | Baseline, at 15 or 60 minutes intervals for 3 hours
  Participants will complete subjective ratings on appetite and well-being
Blood glucose | Baseline, 30, 60, 120 and 180 minutes after breakfast
  Finger prick capillary blood glucose will be collected
Rest of day food record | 8-12 hours
  Parents/guardians will record participants' food intake until the end of the day

CONTACTS AND LOCATIONS:
Overall Officials: Nick Bellissimo, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- School of Nutrition, Ryerson University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided